CLINICAL TRIAL: NCT06028360
Title: The Effect of Virtual Reality (VR) and Progressive Muscle Relaxation (PMR) in Stress Management Among Physiotherapy Students
Brief Title: Progressive Muscle Relaxation (PMR) in Stress Management Among Physiotherapy Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shalamar Institute of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSAHS 2023/02
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Stress
Keywords: Psychological stress; progressive muscle relaxation (PMR)
MeSH Terms: conditions — Stress, Psychological | interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: A Randomized Control Trial with a Control and an Experimental group that will be given intervention 3 consecutive days.
Masking Description: The participants were blind to allocation. They were allocated by simple randomization through lottery method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Muscle Relaxation (Active Comparator): Progressive muscle relaxation will be applied for 15-20 minutes for 3 consecutive days for 1 week.
  Interventions: Other: Progressive Muscle Relaxation
- Virtual Reality (Experimental): Virtual reality session will be given for 8 mins for 3 consecutive days for 1 week.
  Interventions: Other: Progressive Muscle Relaxation; Device: Virtual Reality Therapy

INTERVENTIONS:
Other: Progressive Muscle Relaxation — Intervention will be applied for 15-20 minutes 3 consecutive days a week for 1 week
  Other Names: PMR
Device: Virtual Reality Therapy — Therapy through VR will be given for 8 minutes 3 times a week on consecutively for 1 week
  Other Names: VR Therapy
  Arms: Virtual Reality

SUMMARY:
The objective of this clinical trial is to observe the effect of Virtual Reality (VR) and Progressive muscle relaxation (PMR) in stressed individuals.

Procedure:

Students will be invited verbally and procedure will be explained to them. 20 students will be recruited randomly into control and experimental group. Stress will be predicted using multiple questionnaires. Pss is given before and after the intervention. The students in control group will be given 10 mins session of PMR for 3 consecutive days and in intervention group will be given 10 mins session of PMR followed by 8 mins session of VR for 3 consecutive days in which specific landscapes i.e mountains, forests, nightskies and beaches.

DETAILED DESCRIPTION:
Introduction:

As stress appears to be a natural human response to difficult situations prompting us to address challenges and threats in our lives, prolonged stress may cause the fight or flight response to over-ride body's normal physiology and produce multiple psychological and physiological symptoms resulting in various negative health conditions such as cardiovascular disorders, GIT disturbances, hypertension etc. Moreover, a global survey of adolescents in 72 countries found 66% of students reported feeling stressed about academics and 37% of students felt anxiety relating to schoolwork. Many stress reduction interventions such as Progressive Muscular Relaxation (PMR), mindfulness meditation, deep breathing exercises, and guided imagery have been shown to reduce stress levels among individuals and are being used as traditional relaxation interventions.

Progressive muscle relaxation (PMR) originally known as Jacobson Muscle Relaxation Technique, was developed by Edmund Jacobson in the 1934. It is an actively engaging technique guiding the patients to consciously contract muscles to create tension and release it progressively. This is repeated until patients acquire complete relaxation. Many studies on PMR have proven it to be beneficial in decreasing stress and anxiety levels in many adults as well as children worldwide.

With emerging technology, innovative ideas, such as the use of VR (Virtual Reality) for stress management, have also been considered and studied. According to Cruz-Neira (1993), Virtual reality refers to immersive, interactive, multisensory, viewer-centered, 3D computer generated environments and the combination of technologies required building environments. In the healthcare sector, VR has been proved beneficial for balance and cognition training in cerebral palsy and stroke, and also has been observed to mitigate acute and chronic pain. It can provide rehabilitation, motivation and entertainment all at once. Further studies on its immersive effect suggest it to be helpful in stress management. Natural environments (forests, beaches, mountains etc ) viewed through VR, have shown to help individuals reduce their stress levels, anxiety disorders, and phobias. However, there is little research on individual preferences of different VR landscapes.

In Asia, research relevant to VR has been shown to have a positive effect on stress management in individuals with high stress and mood disorders. Effect of forest and water landscapes on stress management has also been discussed earlier. However, area for more research still remains.

In Pakistan, multiple researches have been conducted on the use of VR in health care and as a rehabilitative intervention for diseases such as stroke, parkinsons, cerebral palsy and amblyopia, but very limited evidence is available on the effect of VR on stress management. No such research has been conducted in this region or in our institution prior to our study.

A study conducted in India showed that the PSS score decreased from mean 22.2 to 16.5 while another study conducted in India indicated that PMR and talk therapy in college students, reduced percieved stress from PSS score of 32.30 to 23.03.

The purpose of our research is to investigate the effect of VR in stress management, the individual preferences of landscapes and its comparison with traditional relaxation technique such as Progressive Muscle Relaxation (PMR). This will help health-care workers improve stress management in a technology driven community.

Statistical analysis:

data will be entered and analyzed using SPSS 25. Numerical data like age, PSS score will be presented in the form of mean ± S.D whereas qualitative data like gender, Pre/Post intervention stress etc. will be presented in the form of Frequency (Percentage). After fulfilling parametric assumptions, Repeated measure ANOVA will be applied.

Potential benefits:

1. The subjects receiving the interventions will experience reduced stress and anxiety.
2. The subjects will be introduced to an innovative and immersive technology i.e., VR.
3. A step will be taken forward towards the use of technology in stress management, along with a traditional relaxation technique such as Progressive muscle relaxation (PMR).
4. The use of VR for stress management is cost effective and time saving.

Potential risks:

1. Motion Sickness It will be tried to minimize by excluding the susceptible subjects, using Visually Induced Motion Sickness Susceptibility Questionnaire (VIMSSQ). Also subjects with any psychological or in-corrected eye sight will not be included in the study. In case the above mentioned risk develops during the intervention, the subject will be given rest.
2. Increased Drop Out Rate If the required sample size is not met due to high drop out rate, new participants will be recruited and the procedure will be repeated until required amount of data is available.

ELIGIBILITY:
Inclusion Criteria:

* Students of either sex, aged between 18-24 years
* Students with Stress (through perceived stress scale PSS, any individual with a score above 14)

Exclusion Criteria:

* Students more susceptible to motion sickness (Through VIMSSQ),
* Students with in-corrected eye-sight,
* Students with phobias relevant to landscapes/views of mountains, forests, beaches and night-skies.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-11-10 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Stress Reduction | the outcome will be determine at the base line of the treatment and at the 3rd day after initiation oftreatment
  Reduction in Perceived Stress scale(PSS) from the previous reading will be considered as stress reduction. information will be collected before and after the treatment on each day. The scoring of Perceived Stress scale(PSS) ranges between 0-40, where 0-13 means low stress, 14-26 means moderate stress and 27-40 would be considered as high perceived stress

CONTACTS AND LOCATIONS:
Overall Officials: Reema Khanam, DPT, Principal Investigator — Shalamar Medical and Dental College; Laiba Khan, DPT, Principal Investigator — Shalamar Medical and Dental College; Maha Sohail, DPT, Principal Investigator — Shalamar Medical and Dental College
Locations (1):
- Shalamar Medical and Dental College, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Gao T, Zhang T, Zhu L, Gao Y, Qiu L. Exploring Psychophysiological Restoration and Individual Preference in the Different Environments Based on Virtual Reality. Int J Environ Res Public Health. 2019 Aug 26;16(17):3102. doi: 10.3390/ijerph16173102. PMID 31455015
- [Background] Wang X, Shi Y, Zhang B, Chiang Y. The Influence of Forest Resting Environments on Stress Using Virtual Reality. Int J Environ Res Public Health. 2019 Sep 5;16(18):3263. doi: 10.3390/ijerph16183263. PMID 31491931
- [Background] Allison S, Irwin Hamilton K, Yuan Y, Wallis Hague G. Assessment of Progressive Muscle Relaxation (PMR) as a Stress-Reducing Technique for First-Year Veterinary Students. J Vet Med Educ. 2020 Dec;47(6):737-744. doi: 10.3138/jvme.2018-0013. Epub 2019 Nov 15. PMID 31738679
- [Background] Ruotolo I, Berardi A, Sellitto G, Panuccio F, Polimeni A, Valente D, Galeoto G. Criterion Validity and Reliability of SF-12 Health Survey Version 2 (SF-12v2) in a Student Population during COVID-19 Pandemic: A Cross-Sectional Study. Depress Res Treat. 2021 Aug 4;2021:6624378. doi: 10.1155/2021/6624378. eCollection 2021. PMID 34394986
- [Background] Levenstein S, Prantera C, Varvo V, Scribano ML, Berto E, Luzi C, Andreoli A. Development of the Perceived Stress Questionnaire: a new tool for psychosomatic research. J Psychosom Res. 1993 Jan;37(1):19-32. doi: 10.1016/0022-3999(93)90120-5. PMID 8421257
- [Background] Keshavarz B, Murovec B, Mohanathas N, Golding JF. The Visually Induced Motion Sickness Susceptibility Questionnaire (VIMSSQ): Estimating Individual Susceptibility to Motion Sickness-Like Symptoms When Using Visual Devices. Hum Factors. 2023 Feb;65(1):107-124. doi: 10.1177/00187208211008687. Epub 2021 Apr 19. PMID 33874752
- [Background] Ahmadpour N, Randall H, Choksi H, Gao A, Vaughan C, Poronnik P. Virtual Reality interventions for acute and chronic pain management. Int J Biochem Cell Biol. 2019 Sep;114:105568. doi: 10.1016/j.biocel.2019.105568. Epub 2019 Jul 12. PMID 31306747
- [Background] Browning MHEM, Shin S, Drong G, McAnirlin O, Gagnon RJ, Ranganathan S, Sindelar K, Hoptman D, Bratman GN, Yuan S, Prabhu VG, Heller W. Daily exposure to virtual nature reduces symptoms of anxiety in college students. Sci Rep. 2023 Jan 23;13(1):1239. doi: 10.1038/s41598-023-28070-9. PMID 36690698
- [Background] Kashif M, Ahmad A, Bandpei MAM, Farooq M, Iram H, E Fatima R. Systematic review of the application of virtual reality to improve balance, gait and motor function in patients with Parkinson's disease. Medicine (Baltimore). 2022 Aug 5;101(31):e29212. doi: 10.1097/MD.0000000000029212. PMID 35945738